CLINICAL TRIAL: NCT01151358
Title: Multicenter Prospective Evaluation of Patient- and Lesion Specific Prognostic Factors for Standard RadioImmunoTherapy With 90-Yttrium-labeled Anti-CD20 in Follicular Non-Hodgkin´s Lymphoma
Brief Title: Evaluation of Patient and Lesion Specific Prognostic Factors for Standard Radioimmunotherapy
Acronym: MERIT-NHL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Saarland (Other)
Responsible Party: Carl-Martin Kirsch, MD, University Hospital, Saarland
Other Study IDs: MERIT-NHL
Record Dates: First submitted 2010-06-24; First posted 2010-06-28 (Estimated); Last update posted 2010-06-28 (Estimated); Status verified 2010-06

CONDITIONS: Follicular Lymphoma
Keywords: radioimmunotherapy; follicular non-Hodgkin´s lymphoma; FDG-PET; prognostic factors; multicenter study
MeSH Terms: conditions — Lymphoma, Follicular

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
MERIT-NHL as an addendum to the International Registry of Radioimmunotherapy (RIT registry) pooling clinical data of patients who suffered from a non-Hodgkin´s lymphoma also includes the documentation of the respective FDG-PET and CT-image files in an online archive.

Based on these documented clinical and imaging data, the MERIT study group centrally performs an intra- as well as interindividual evaluation of follicular CD20+ lymphoma lesions before and after radioimmunotherapy. According to this, the aim of the MERIT-NHL study is to prospectively identify yet unknown patient- and lesion specific prognostic factors predicting patient´s outcome in line with the therapeutic modality radioimmunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* standard radioimmunotherapy with 90-yttrium-labeled anti-CD20-antibodies in treatment of relapsed and/or refractory follicular NHL or partial remission after induction chemotherapy
* finding of at least one image-guided measurable lymphoma lesion
* existence of FDG-PET- and CT-image data of at most 8 weeks before treatment
* signed patient´s agreement for RIT registry and MERIT-NHL

Exclusion Criteria:

* other therapy modalities than standard radioimmunotherapy (e.g. consolidation)
* solely CNS-lymphoma or primary effusion lymphoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who suffer from a relapsed and/or refractory follicular non-Hodgkin´s lymphoma (FL) or patients with partial remission after induction chemotherapy of FL
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2008-05; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of patient- and lesion specific prognostic factors of radioimmunotherapy | 3 years

SECONDARY OUTCOMES:
Detection of diagnostical relevance of FDG-PET- and CT-image data findings in staging and re-staging of follicular non-Hodgkin´s lymphoma as well as in documentation of patient´s outcome after standard radioimmunotherapy | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Carl-Martin Kirsch, MD, Principal Investigator — Universitaetsklinikum des Saarlandes
Locations (4):
- Germany (4):
  - Dept. of Nuclear Medicine, Saarland University Hospital, Homburg (Saar), Saarland
  - Klinikum Karlsruhe, Dept. of Nuclear Medicine, Karlsruhe
  - University Clinic Kiel-Luebeck, Lübeck
  - Technical University, Dept. of Nuclear Medicine, Munich